CLINICAL TRIAL: NCT04281966
Title: Testing the Efficacy of the Ability School Engagement Partnership Program (ASEP)
Acronym: ASEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Queensland (Other)
Collaborators: Restorative Outcomes Australia (Unknown); Department of Education, Queensland (Unknown); Queensland Police Service (Unknown); Australian Department of Social Services (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019002851
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: School Attendance; Welfare Dependence; Antisocial Behavior
Keywords: School Attendance; Welfare Dependence; Antisocial Behavior; Third-Party Policing Partnerships
MeSH Terms: conditions — Antisocial Personality Disorder

STUDY DESIGN:
Intervention Model Description: The current project utilizes a randomized controlled cluster trial to assess the efficacy of the ASEP intervention and thereby theoretically test the efficacy of third-party-policing. Data will be collected from high schools that are in either socially disadvantaged areas or have students who reside in socially disadvantaged areas. A total of 69 high schools were identified as eligible for the Trial based upon measures of social disadvantage. The 69 eligible high schools were randomly assigned to participate in the ASEP (experiment) or business-as-usual (control) conditions. Young people from schools who take part in the ASEP (experiment) will be recruited from the experimental schools. Official data will be obtained about the young people (identified for those in the experimental condition who consent; de-identified for the young people in the control schools).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment (Experimental): For young people from schools randomly assigned to the experimental ASEP condition will participate in the ASEP intervention. The ASEP intervention is a Third-Party Policing partnership that involves a partnership between police and school, an ASEP conference and follow up which is organized and led by a conference facilitator with the young person, their parent (or guardian), a school representative (e.g., teacher), and a uniformed school-based police officer. The police and school representatives will be trained by the facilitator to utilize procedurally just dialogue during the entirety of the conference. The ASEP conference script will utilize a procedurally just dialogue to increase both the young person and their parents' perceptions and knowledge of the legitimacy of the truancy laws, police, and schools in order to gain willing compliance to follow the rules.
  Interventions: Behavioral: Ability School Engagement Program Conference
- Control (No Intervention): Participants allocated to the control condition will be given the "business-as-usual' approach to handling school non-attendance. The control participants will be sanctioned in the usual manner for engaging in truancy through the requirements denoted in the Queensland Education (General Provisions) Act (2006).

INTERVENTIONS:
Behavioral: Ability School Engagement Program Conference — The ASEP conference focuses on understanding the reasons behind why the young person is not attending school regularly, understand how the young person's non-attendance affects other conference participants, highlight the legal consequences of parents and/or guardians to ensure that their child attends school, and the development of a young person-centered Action Plan, which will specifically detail the "actions" that all parties are to take over the next three months to ensure that the young person re-engages with school and/or transitions into paid work.
  Arms: Experiment

SUMMARY:
This project is an up-scaled test of the Ability School Engagement Partnership (ASEP) Project. The ASEP is a partnership program that aims to increase school attendance and is grounded in the theory of Third-Party-Policing (TPP). In ASEP, school-based police officers partner with schools (i.e., the third-party) who have legal powers to control and prevent school absenteeism. The ASEP intervention includes an ASEP conference in which the legal requirements to attend school are explicitly communicated in a procedurally just way to young people missing school and their parents/guardians. Restorative Outcomes Australia (ROA) is a provide provider partner who will oversee the facilitation of the ASEP conferences. While the program is designed to re-engage these young people in school and/or facilitate transitions to work and reduce antisocial behavior (e.g., delinquency), this trial will also test the capacity of the program to improve collaboration between the schools and police and also monitor young participants' future life outcomes, such as future welfare dependence.

DETAILED DESCRIPTION:
The ASEP is grounded in the theory of Third Party Policing (TPP). TPP interventions focus on controlling negative behavioral outcomes through partnerships that use a third party's legal powers. In ASEP, the police partner with the schools to work together to engage with young people, reduce their anti-social behavior and increase their school attendance. At the core of the partnership is communication of the legal lever: in ASEP, it is the Queensland Education (General Provisions) Act (2006) - requiring young people attend school up to age 16 and holding parents legally responsible. The laws are communicated to parents and young people who are not regularly attending school in a procedurally fair way within the context of an ASEP conference. The ASEP conference is especially designed to incorporate fair communication of the laws and consequences and involves a purpose-built script that seeks to increase willingness of both parents and young people to comply with the law. The ASEP conference participants include a trained facilitator (from Restorative Outcomes Australia; ROA), the young person missing a lot of school, their parent or guardian, a uniformed school-based police officer, and a school representative (e.g., teacher). An individually tailored Action Plan is developed during the conference which stipulate the "actions" that all conference participants are to take over the subsequent two months in order to ensure that the young person increases their school attendance and re-engages with school and/or transitions into paid work.

ELIGIBILITY:
Inclusion Criteria:

* High school aged young people only, aged 12 to 16;
* Have 15% or more unexplained absences over each other previous two school terms;
* Have no known legitimate explanation for absences (e.g., ongoing medical issue); and
* Have at least one responsibly adult in their lives (e.g., parent, guardian, or carer) who provides social and/or financial support.

Exclusion Criteria:

* None

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 753 (Estimated)
Dates: Start 2019-06-21 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Official School Absences | Six-Months Post-Intervention
  A count of the number of school absences of young people.
Official Arrest Records | Six-Months Post Intervention
  A count of official arrest records of young people.
Perceptions of School Legitimacy | Two-months post intervention
  These measures are adapted from the original ASEP Project Trial (Mazerolle, 2014). The original ASEP researchers adapted these scales from Murphy and Mearns (2008), Sunshine and Tyler (2003), and Tankebe (2009). These indices include five items that address respondents' (young people and parents/guardians in the experimental group only) perceptions of legitimacy of school staff with higher values equating to better perceptions of school staff legitimacy.
Perceptions of School Procedural Justice | Two-months post intervention
  These measures are adapted from the original ASEP Project Trial (Mazerolle, 2014). The original ASEP researchers adapted these scales from Murphy and Mearns (2008), Sunshine and Tyler (2003), and Tankebe (2009). These indices include five items that address respondents' (young people and parents/guardians in the experimental group only) perceptions of procedural justice of school staff with higher values equating to better perceptions of school staff procedural justice.
Perceptions of Police Legitimacy | Two-months post intervention
  These measures are adapted from the original ASEP Project Trial (Mazerolle, 2014). The original ASEP researchers adapted these scales from Murphy and Mearns (2008), Sunshine and Tyler (2003), and Tankebe (2009). These indices include five items that address respondents' (young people and parents/guardians in the experimental group only) perceptions of legitimacy of police in general with higher values equating to better perceptions of police legitimacy.
Perceptions of Police Procedural Justice | Two-months post intervention
  These measures are adapted from the original ASEP Project Trial (Mazerolle, 2014). The original ASEP researchers adapted these scales from Murphy and Mearns (2008), Sunshine and Tyler (2003), and Tankebe (2009). These indices include five items that address respondents' (young people and parents/guardians in the experimental group only) perceptions of procedural justice of police in general.
Perceptions of Family Legitimacy | Two-months post intervention
  Adapted from the work of Trinkner, 2012; Trinkner et al., 2012; Trinker & Cohn, 2014. Measures respondents' (young people and parents/guardians in the experimental group only) perceptions of family legitimacy with higher values equating to better perceptions of family legitimacy.
Perceptions of Family Procedural Justice | Two-months post intervention
  Adapted from the work of Trinkner, 2012; Trinkner et al., 2012; Trinker & Cohn, 2014. Measures respondents' (young people and parents/guardians in the experimental group only) perceptions of family procedural justice with higher values equating to better perceptions of family legitimacy.
General Well-being | Two-months post intervention
  The Short Warwick-Edinburgh Mental Well-being Scale (SWEMWBS; Haver et al., 2015; Stewart-Brown et al., 2009; Taggart et al., 2015; Tennant et al., 2007) to be administered to young people and parents in the experimental condition only. It includes 7 items, scores range from 7 to 35, and higher scores coincide with better well-being.
Self-efficacy | Two-months post intervention
  Includes 12 items from the Coping Orientation to Problems Experienced (COPE) Inventory (Carver et al., 1989; Carver, 1997) to be administered to young people and parents in the experimental condition only. Scores will range from 12 to 48 and coded so that higher values equate to better coping skills.

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine Mazerolle, Ph.D., Principal Investigator — The University of Queensland; Sarah Bennett, Ph.D., Principal Investigator — The University of Queensland; Stephanie Cardwell, Ph.D., Principal Investigator — The University of Queensland
Locations (1):
- The University of Queensland, Brisbane, Queensland, Australia

REFERENCES:
- [Background] Antrobus, E., Bennett, S., Mazerolle, L., & Eggins, E. (2019). Parental and student perceptions of procedural justice and legitimacy in the context of truancy: Results from a randomized field trial. Australian & New Zealand Journal of Criminology, 52(4), 534-557.
- [Background] Bennett, S., Mazerolle, L., Antrobus, E., Eggins, E., & Piquero, A. R. (2018). Truancy intervention reduces crime: Results from a randomized field trial. Justice Quarterly, 35(2), 309-329.
- [Background] Cardwell, S. M., Mazerolle, L., & Piquero, A. R. (2019). Parental attachment and truant rationalizations of antisocial behavior: findings from a randomized controlled trial. Journal of Crime and Justice, 1-19.
- [Background] Cardwell, S. M., Mazerolle, L., & Piquero, A. R. (2019). Truancy intervention and violent offending: Evidence from a randomized controlled trial. Aggression and Violent Behavior, 49.
- [Background] Cardwell, S. M., Mazerolle, L., Bennett, S., & Piquero, A. R. (2019). Changing the relationship between impulsivity and antisocial behavior: the impact of a school engagement program. Crime & Delinquency, 65(8), 1076-1101.
- [Background] Carver CS, Scheier MF, Weintraub JK. Assessing coping strategies: a theoretically based approach. J Pers Soc Psychol. 1989 Feb;56(2):267-83. doi: 10.1037//0022-3514.56.2.267. PMID 2926629
- [Background] Cohn, E. S., Trinkner, R. J., Rebellon, C. J., Van Gundy, K. T., & Cole, L. M. (2012). Legal attitudes and legitimacy: Extending the integrated legal socialization model. Victims & Offenders, 7(4), 385-406.
- [Background] Mazerolle, L. (2014). The power of policing partnerships: Sustaining the gains. Journal of Experimental Criminology, 10(3), 341-365.
- [Background] Mazerolle L, Antrobus E, Bennett S, Eggins E. Reducing Truancy and Fostering a Willingness to Attend School: Results from a Randomized Trial of a Police-School Partnership Program. Prev Sci. 2017 May;18(4):469-480. doi: 10.1007/s11121-017-0771-7. PMID 28317075
- [Background] Mazerolle, L., Antrobus, E., Cardwell, S. M., Piquero, A. R., & Bennett, S. (2019). Harmonizing legal socialization to reduce antisocial behavior: Results from a randomized field trial of truanting young people. Justice Quarterly, 1-28.
- [Background] Mazerolle, L., Bennett, S., Antrobus, E., Cardwell, S. M., Eggins, E., & Piquero, A. R. (2019). Disrupting the pathway from truancy to delinquency: a randomized field trial test of the longitudinal impact of a school engagement program. Journal of Quantitative Criminology, 35(4), 663-689.
- [Background] Murphy, K., & Mearns, M. (2008). The Public Safety and Security in Australia Survey: Survey methodology and preliminary findings. ARC Centre for Excellence in Policing and Security (Working Paper, October 2008). The Australian National University.
- [Background] Sunshine, J., & Tyler, T. R. (2003). The role of procedural justice and legitimacy in shaping public support for policing. Law & Society Review, 37(3), 513-548.
- [Background] Tankebe, J. (2009). Public cooperation with the police in Ghana: Does procedural fairness matter? Criminology, 47(4), 1265-1293.
- [Background] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300
- [Background] Trinkner, R. (2012). Testing the procedural justice model of legal socialization: Expanding beyond the legal world. (Doctoral dissertation). University of New Hampshire, Durham, New Hampshire.
- [Background] Trinkner R, Cohn ES, Rebellon CJ, Van Gundy K. Don't trust anyone over 30: parental legitimacy as a mediator between parenting style and changes in delinquent behavior over time. J Adolesc. 2012 Feb;35(1):119-32. doi: 10.1016/j.adolescence.2011.05.003. Epub 2011 Jun 12. PMID 21669454
- [Background] Trinkner R, Cohn ES. Putting the "social" back in legal socialization: procedural justice, legitimacy, and cynicism in legal and nonlegal authorities. Law Hum Behav. 2014 Dec;38(6):602-17. doi: 10.1037/lhb0000107. Epub 2014 Sep 22. PMID 25243981
- [Background] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744
- [Background] Haver A, Akerjordet K, Caputi P, Furunes T, Magee C. Measuring mental well-being: A validation of the Short Warwick-Edinburgh Mental Well-Being Scale in Norwegian and Swedish. Scand J Public Health. 2015 Nov;43(7):721-7. doi: 10.1177/1403494815588862. Epub 2015 Jun 3. PMID 26041133
- [Background] Stewart-Brown S, Tennant A, Tennant R, Platt S, Parkinson J, Weich S. Internal construct validity of the Warwick-Edinburgh Mental Well-being Scale (WEMWBS): a Rasch analysis using data from the Scottish Health Education Population Survey. Health Qual Life Outcomes. 2009 Feb 19;7:15. doi: 10.1186/1477-7525-7-15. PMID 19228398
- [Background] Taggart, F., Stewart-Brown, S., & Parkinson, J. (2015). Warwick-Edinburgh Mental Well-being Scale (WEMWBS) User Guide, Version 2. NHS Health Scotland.
- See also: Crime Solutions: Ability School Engagement Program — https://www.crimesolutions.gov/ProgramDetails.aspx?ID=580